CLINICAL TRIAL: NCT03674541
Title: The Exercise Response to Pharmacologic Cholinergic Stimulation in Myalgic Encephalomyelitis / Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Systrom, Principal Investigator; Director, Dyspnea Center; Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018P001871
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome; Chronic Fatigue Syndrome; Myalgic Encephalomyelitis; Exercise Intolerance; Dysautonomia; Low Ventricular Filling Pressures (Preload Failure); Postural Orthostatic Tachycardia Syndrome; Orthostatic Hypotension; Fibromyalgia
Keywords: Myalgic encephalomyelitis/Chronic fatigue syndrome; Myalgic encephalomyelitis; Chronic fatigue syndrome; Pyridostigmine; Exercise Intolerance; Invasive Cardiopulmonary Exercise Test
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Autonomic Nervous System Diseases; Postural Orthostatic Tachycardia Syndrome; Hypotension, Orthostatic; Fibromyalgia | interventions — Pyridostigmine Bromide; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned randomly to receive either pyridostigmine or placebo, both study participants and investigators will be blinded.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Drug - Pyridostigmine (Active Comparator): Pyridostigmine 60 mg by mouth as a one time dose
  Interventions: Drug: Pyridostigmine Bromide
- Placebo (Placebo Comparator): Placebo by mouth as a one time dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine Bromide — Pyridostigmine Bromide 60 mg capsule by mouth as a one time dose
  Other Names: Mestinon
  Arms: Study Drug - Pyridostigmine
Drug: Placebo — Placebo (Cellulose microcrystalline) capsule by mouth as a one time dose
  Other Names: Cellulose microcrystalline
  Arms: Placebo

SUMMARY:
Myalgic encephalomyelitis/Chronic fatigue syndrome (ME/CFS), otherwise known as Chronic fatigue syndrome (CFS) or myalgic encephalomyelitis (ME), is an under-recognized disorder whose cause is not yet understood. Suggested theories behind the pathophysiology of this condition include autoimmune causes, an inciting viral illness, and a dysfunctional autonomic nervous system caused by a small fiber polyneuropathy. Symptoms include fatigue, cognitive impairments, gastrointestinal changes, exertional dyspnea, and post-exertional malaise. The latter two symptoms are caused in part by abnormal cardiopulmonary hemodynamics during exercise thought to be due to a small fiber polyneuropathy. This manifests as low biventricular filling pressures throughout exercise seen in patients undergoing an invasive cardiopulmonary exercise test (iCPET) along with small nerve fiber atrophy seen on skin biopsy.

After diagnosis, patients are often treated with pyridostigmine (off-label use of this medication) to enhance cholinergic stimulation of norepinephrine release at the post-ganglionic synapse. This is thought to improve venoconstriction at the site of exercising muscles, leading to improved return of blood to the heart and increasing filling of the heart to more appropriate levels during peak exercise. Retrospective studies have shown that noninvasive measurements of exercise capacity, such as oxygen uptake, end-tidal carbon dioxide, and ventilatory efficiency, improve after treatment with pyridostigmine. To date, there are no studies that assess invasive hemodynamics after pyridostigmine administration.

It is estimated that four million people suffer from ME/CFS worldwide, a number that is thought to be a gross underestimate of disease prevalence. However, despite its potential for debilitating symptoms, loss of productivity, and worldwide burden, the pathophysiology behind ME/CFS remains unknown and its treatment unclear. By evaluating the exercise response to cholinergic stimulation, this study will shed further light on the link between the autonomic nervous system and cardiopulmonary hemodynamics, potentially leading to new therapeutic targets.

DETAILED DESCRIPTION:
The hypothesis of our study is that hemodynamic, ventilatory and oxygen exchange variables such biventricular filling pressures and systemic oxygen extraction can be improved by cholinergic stimulation in patients with ME/CFS.

The objective of this study is to examine the exercise response to pharmacologic cholinergic stimulation in ME/CFS patients already undergoing a clinically indicated invasive cardiopulmonary exercise test (iCPET). This will be achieved by inhibiting acetylcholinesterase with pyridostigmine, thus increasing acetylcholine levels, downstream levels of norepinephrine, and enhancing vascular regulation.

To test our hypothesis, we propose the following specific aims:

Define the response of peak oxygen uptake(VO2) to pyridostigmine. Define the gas exchange responses, such as end-tidal carbon dioxide(CO2) and ventilatory efficiency to pyridostigmine.

Define the hemodynamic responses, such as right atrial pressures, pulmonary artery pressure, pulmonary capillary wedge pressures, cardiac output, heart rate, stroke volume, pulmonary vascular resistance and systemic vascular resistance to pyridostigmine.

Evaluate the response of skeletal muscle oxygen extraction and lactate to pyridostigmine.

These determinations will occur during a clinically indicated iCPET, which includes exercising on a stationary cycle with a right heart catheter (RHC) and a radial arterial line in place. To stimulate the cholinergic response, a single dose of an oral acetylcholinesterase inhibitor, pyridostigmine, versus placebo will be given after the iCPET. Recovery cycling will be performed after a rest period of 50 minutes. This will be administered in a randomized, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Institute of Medicine (IOM) criteria for ME/CFS
* Completing the clinically indicated invasive cardiopulmonary exercise test (iCPET)

Exclusion Criteria:

* Obesity (BMI > 30 kg/m2)
* Non-controlled asthma
* Anemia (Hb < 10 g/dl)
* Active or treated cancer
* History of interstitial lung disease (ILD)
* Chronic obstructive pulmonary disease (COPD)
* Pulmonary hypertension (PH)
* Congestive heart failure (CHF)
* Active arrhythmias
* Valvular heart disease
* Coronary artery disease (CAD)
* Other conditions that could predict a limitation or not completion of the study.
* Pregnancy
* Submaximal testing in clinically indicated iCPET
* Pulmonary mechanical limitation to exercise in clinically indicated iCPET.
* Pulmonary arterial hypertension in clinically indicated iCPET.
* Pulmonary venous hypertension in clinically indicated iCPET.
* Exercise induced pulmonary arterial hypertension in clinically indicated iCPET.
* Exercise induced pulmonary venous hypertension in clinically indicated iCPET.
* Persistent hypotension during or after the clinically indicated iCPET.
* Refractory arrhythmia during or after the clinically indicated level 3 CPET.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Systrom, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification(text, tables, figures, and appendices) will be available for researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to jsquires1@bwh.harvard.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Joseph P, Pari R, Miller S, Warren A, Stovall MC, Squires J, Chang CJ, Xiao W, Waxman AB, Systrom DM. Neurovascular Dysregulation and Acute Exercise Intolerance in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Randomized, Placebo-Controlled Trial of Pyridostigmine. Chest. 2022 Nov;162(5):1116-1126. doi: 10.1016/j.chest.2022.04.146. Epub 2022 May 6. PMID 35526605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from PI's clinic
Period: Overall Study
Arm/Group | Study Drug - Pyridostigmine | Placebo
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Groups:
- Placebo (Female): Placebo by mouth as a one time dose
  Placebo: Placebo (Cellulose microcrystalline) capsule by mouth as a one time dose
- Placebo (Male): Placebo by mouth as a one time dose
  Placebo: Placebo (Cellulose microcrystalline) capsule by mouth as a one time dose
  Not included in statistical analysis
- Total: Total of all reporting groups
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male) | Total
Number analyzed (Participants) | 23 | 16 | 6 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40 (16) | 40 (11) | 50 (20) | 42 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 0 | 39
  Male | 0 | 0 | 6 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 12 | 4 | 37
  Other | 2 | 4 | 2 | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.8 (2.7) | 23.0 (4.1) | 23.8 (2.7) | 23.5 (3.3)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.9 (1.3) | 14.0 (1.1) | 15.7 (1.4) | 14.2 (1.3)
Hypertension [Count of Participants; unit: Participants] | 3 | 1 | 1 | 5
Dyslipidemia [Count of Participants; unit: Participants] | 1 | 1 | 2 | 4
Obesity [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Cardiovascular Family History [Count of Participants; unit: Participants] | 13 | 11 | 2 | 26
Diabetes Mellitus [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Previous Myocardial Infarction [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Coronary Artery Disease [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Statins [Count of Participants; unit: Participants] | 2 | 0 | 2 | 4
Beta Blockers [Count of Participants; unit: Participants] | 2 | 1 | 0 | 3
Acetylsalicylic Acid [Count of Participants; unit: Participants] | 2 | 0 | 0 | 2
Calcium Channel Blockers [Count of Participants; unit: Participants] | 1 | 0 | 0 | 1
Diuretics [Count of Participants; unit: Participants] | 1 | 0 | 2 | 3
Angiotensin-converting enzyme (ACE) Inhibitors [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Objective Evidence of small fiber neuropathy by Morphological and/or Functional Testing [Count of Participants; unit: Participants] — Population: Not all participants underwent morphological and/or functional testing for small fiber neuropathy (SFN)
  Participants
    number analyzed (Participants) | 22 | 15 | 3 | 40
    (all) | 11 | 3 | 0 | 14
Epidermal Skin Biopsy Evidence of SFN [Count of Participants; unit: Participants] — Population: Not all participants underwent epidermal skin biopsies for small fiber neuropathy (SFN)
  Participants
    number analyzed (Participants) | 21 | 15 | 3 | 39
    (all) | 5 | 2 | 0 | 7
Sweat Gland Biopsy Evidence of SFN [Count of Participants; unit: Participants] — Population: Not all participants underwent sweat gland biopsies for small fiber neuropathy (SFN)
  Participants
    number analyzed (Participants) | 8 | 4 | 3 | 15
    (all) | 5 | 0 | 0 | 5
Functional Testing (QSART and/or ESC) Evidence of SFN [Count of Participants; unit: Participants] — Population: Not all participants underwent functional testing (QSART and/or ESC) for small fiber neuropathy (SFN)
  Participants
    number analyzed (Participants) | 10 | 6 | 3 | 19
    (all) | 1 | 1 | 0 | 2
POTS (Postural Orthostatic Tachycardia Syndrome) [Count of Participants; unit: Participants] | 13 | 5 | 1 | 19
Fibromyalgia [Count of Participants; unit: Participants] | 6 | 5 | 3 | 14
Mast Cell Activation Syndrome [Count of Participants; unit: Participants] | 4 | 3 | 0 | 7
Preceding Infection [Count of Participants; unit: Participants] | 12 | 8 | 4 | 24
Positive Antinuclear Antibody [Count of Participants; unit: Participants] | 7 | 3 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Uptake (Peak VO2) Between the First and Second iCPET
Description: Define the response of oxygen uptake to pyridostigmine expressed both as mL/min and mL/min/kg. The difference in peak oxygen uptake from first iCPET to second iCPET. Research has shown that ME/CFS patients have inability to reproduce results on two consecutive cardiopulmonary exercise tests(CPET). Traditionally this is demonstrated with a two-day CPET protocol, but in this study we investigate the acute effects of pyridostigmine administration on the early stages of post exertional malaise(PEM).
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
mL/min | 13.3 (13.4) | -40.3 (21.3) | 111.8 (65.0)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.043, Welch's t-test

2. Secondary Outcome: Peak-Rest Oxygen Uptake (VO2)
Description: Peak versus rest changes in oxygen uptake between first and second CPETs expressed as mL/min.
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
mL/min | 25.9 (15.3) | -60.8 (25.6) | 121.8 (80.0)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.008, Welch's t-test — P-value was not adjusted for multiplicity for secondary outcomes

3. Secondary Outcome: Peak Cardiac Output (Qc)
Description: Arterial and mixed-venous blood gases and pH are measured at peak exercise and Qc is calculated using the direct Fick principle Qc=VO2/(Ca-Cv). Change in peak Qc between first and second iCPETs is measured in L/min.
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
L/min | 0.2 (0.2) | -0.2 (0.3) | 1.1 (0.4)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.263, Welch's t-test — Not adjusted for multiplicity

4. Secondary Outcome: Peak-Rest Cardiac Output (Qc)
Description: Peak versus rest change in cardiac output expressed in L/min between first and second iCPETs. Cardiac output is determined using the direct Fick principle.
Time Frame: First iCPET up to 30 min, 50 minutes rest, second iCPET up to 30 minutes
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
L/min | -0.2 (0.6) | -1.9 (0.6) | 0.9 (0.8)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.039, Welch's t-test — Not adjusted for multiplicity

5. Secondary Outcome: Peak Right Atrial Pressure (RAP)
Description: Difference in peak RAP between first and second iCPETs measured in mmHg.
Time Frame: First iCPEt up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
mm Hg | 1.2 (0.3) | 0.1 (0.5) | 1.7 (0.7)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.068, Welch's t-test — Not adjusted for multiplicity

6. Secondary Outcome: Peak-Rest Right Atrial Pressure (RAP)
Description: Peak versus rest changes in RAP between first and second iCPETs measured in mmHg
Time Frame: First iCPEt up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
mm Hg | 1.0 (0.5) | -0.6 (0.5) | 0.0 (1.0)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.045, Welch's t-test — Not adjusted for multiplicity

7. Secondary Outcome: Peak Pulmonary Arterial Wedge Pressure (PAWP)
Description: Difference in peak PAWP between first and second iCPETs measured in mmHg
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
mm Hg | 1.0 (0.8) | 1.0 (0.5) | 1.5 (1.4)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 1.000, Welch's t-test — Not adjusted multiplicity

8. Secondary Outcome: Peak Stroke Volume (SV)
Description: Difference in peak SV between first and second iCPETs measured in mL
Time Frame: First iCPEt up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: mL
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
mL | 3.0 (1.4) | -1.1 (1.9) | -12.7 (12.9)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.093, Welch's t-test — Not adjusted for multiplicity

9. Secondary Outcome: Peak (Ca-vO2)/[Hgb]
Description: Difference in peak arterial-venous oxygen content difference normalized to hemoglobin (Ca-vO2)/[Hgb] between first and second iCPETs
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 5
Ratio | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.1)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.427, Welch's t-test — Not adjusted for multiplicity

10. Secondary Outcome: Ventilatory Efficiency (VE/VCO2)
Description: Difference in ventilatory efficiency between first and second iCPETs
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
Ratio | -0.2 (0.8) | 1.0 (0.6) | 1.7 (0.6)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.262, Welch's t-test — Not adjusted for multiplicity

11. Secondary Outcome: Borg Fatigue Scale
Description: Difference in perception of fatigue at peak exercise between first and second iCPETs. Used Borg Scale 0 (minimal) to 10 (maximal).
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
units on a scale | 0.1 (0.2) | -0.6 (0.3) | 0.4 (0.4)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.038, Welch's t-test — Not adjusted for multiplicity

12. Secondary Outcome: Borg Dyspnea Scale
Description: Difference in perceived dyspnea at peak exercise between first and second iCPETs. Used Borg Scale 0 (minimal) to 10 (maximal).
Time Frame: First iCPET up to 30 minutes, 50 minutes rest, second iCPET up to 30 minutes.
Population: Data was collected for all 45 patient, 23 females on study drug, 22 on placebo (16 females, 6 males).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Study Drug - Pyridostigmine | Placebo (Female) | Placebo (Male)
Number analyzed (Participants) | 23 | 16 | 6
units on a scale | -0.1 (0.2) | -1.0 (0.5) | 0.3 (0.5)
Statistical Analysis 1: Comparison: Study Drug - Pyridostigmine vs Placebo (Female); Test type: Superiority; p = 0.147, Welch's t-test

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the two iCPETs and for the duration of the 50 minutes rest between the two iCPETs. After the second iCPET, the subjects were monitored for an hour in the recovery room. The subjects received a follow up phone call or email up to one week following the day of the procedure to assess if they experienced any adverse events from the study. This was documented for every patient.
Description: Collection of adverse events after subject had been discharged from the site was based on a follow-up phone call or email up to one week following the day of the iCPET.
Groups:
- Placebo: Placebo by mouth as a one time dose
  Placebo: Placebo (Cellulose microcrystalline) capsule by mouth as a one time dose
  Deaths and Adverse Events for the Placebo Arm were collected together regardless of sex
Arm/Group | Study Drug - Pyridostigmine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 15/23 | 15/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Drug - Pyridostigmine (N=23) | Placebo (N=22)
Post-Exertional Malaise (PEM) (Immune system disorders) | 13 | 11 — Hallmark of ME/CFS. Manifestation of flu-like symptoms following physical or emotional exertion.
Wrist Pain (Skin and subcutaneous tissue disorders) | 2 | 4 — Residual pain from catheterization of radial artery

LIMITATIONS AND CAVEATS:
Of the 45 subjects, 39 were female and 6 were male. Although this gender distribution is reflective of the gender differences seen in ME/CFS, our small sample size produced a randomization error where all 6 male participants were placed in the placebo group. We elected not to include males in the statistical analysis as their response to exercise was discordant compared to females who received placebo. In addition, reducing the sample size increases the likelihood of type II errors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT03674541/Prot_SAP_000.pdf